CLINICAL TRIAL: NCT01563471
Title: Single-centre, Randomised, Placebo-controlled, Double-blind, Dose Escalation Trial Investigating Pharmacokinetics, Pharmacodynamics and Tolerability of Three Different Single Intravenous Doses of Activated Recombinant Factor VIIa (rFVIIa/NovoSeven®) in Healthy Caucasian and Japanese Subjects
Brief Title: Safety and Tolerability of Intravenous Doses of Activated Recombinant Human Factor VII in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: F7LIVER-1465
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors; Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment sequence 1 (Experimental)
  Interventions: Drug: activated recombinant human factor VII; Drug: placebo
- Treatment sequence 2 (Experimental)
  Interventions: Drug: activated recombinant human factor VII; Drug: placebo
- Treatment sequence 3 (Experimental)
  Interventions: Drug: activated recombinant human factor VII; Drug: placebo
- Treatment sequence 4 (Placebo Comparator)
  Interventions: Drug: activated recombinant human factor VII; Drug: placebo

INTERVENTIONS:
Drug: activated recombinant human factor VII — Subjects will be randomised to one of four treatment sequences. Subjects will receive single bolus i.v. injection of 40, 80 or 160 mcg/kg body weight of trial drug or placebo on each day of the three separate visits
Drug: placebo — Subjects will be randomised to one of four treatment sequences. Subjects will receive single bolus i.v. injection of 40, 80 or 160 mcg/kg body weight of trial drug or placebo on each day of the three separate visits

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the pharmacokinetics of three different single doses activated recombinant human factor VII in Caucasian and Japanese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian or Japanese
* Healthy as defined by medical history, physical and biological examinations

Exclusion Criteria:

* History of allergy or hypersensitivity reaction to any medication
* History or presence of any organic disorder likely to modify absorption, distribution or elimination of the medication
* Alcohol or substance abuse disorder
* Subject in his exclusion period in the Healthy Volunteers National Register of the French Ministry of Health

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2001-10; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Area under the Curve (AUC) of FVII:C (Factor VII clotting activity) from 0-24 hours

SECONDARY OUTCOMES:
Mean residence time (MRT)
Maximum plasma concentration (Cmax)
Time to reach maximum plasma concentration (tmax)
Area under the Curve (AUC) from 0-24 hours of the PT (Prothrombin Time)
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Paris, France

REFERENCES:
- [Result] Fridberg MJ, Hedner U, Roberts HR, Erhardtsen E. A study of the pharmacokinetics and safety of recombinant activated factor VII in healthy Caucasian and Japanese subjects. Blood Coagul Fibrinolysis. 2005 Jun;16(4):259-66. doi: 10.1097/01.mbc.0000169218.15926.34. PMID 15870545
- [Result] Levy JH, Fingerhut A, Brott T, Langbakke IH, Erhardtsen E, Porte RJ. Recombinant factor VIIa in patients with coagulopathy secondary to anticoagulant therapy, cirrhosis, or severe traumatic injury: review of safety profile. Transfusion. 2006 Jun;46(6):919-33. doi: 10.1111/j.1537-2995.2006.00824.x. PMID 16734808
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com